CLINICAL TRIAL: NCT05328674
Title: Clinical and Comparative Evaluation of the Treatment Results of Arthroscopic Reconstruction of Cartilage Defects in the Knee Joint With the Use of Autogenous Cartilage Graft With PRP GF (Platelet-rich Plasma With Growth Factors).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: eMKa MED Medical Center (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-563/2021
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-03

CONDITIONS: Cartilage Damage; Cartilage Injury; Knee Injuries
Keywords: Cartilage; Injury; Damage; Defects; Techniques; Reconstruction
MeSH Terms: conditions — Knee Injuries; Wounds and Injuries | interventions — Intercellular Signaling Peptides and Proteins

STUDY DESIGN:
Intervention Model Description: comparison of the results of arthroscopic treatment of analogous areas of cartilage defects in the knee joint obtained in study groups using two methods: microfracture and autogenous PRP GF cartilage graft (Auto Cart - Arthrex method).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfracture method (Active Comparator)
  Interventions: Procedure: Arthroscopic reconstruction of the cartilage defects of the knee joint using the microfracture method
- Method of autogenous PRP (Auto Cart-Arthrex) cartilage transplant (Experimental)
  Interventions: Procedure: Arthroscopic reconstruction of cartilage defects in the knee joint with the use of autogenous cartilage transplant with PRP GF (platelet plasma with growth factor)

INTERVENTIONS:
Procedure: Arthroscopic reconstruction of cartilage defects in the knee joint with the use of autogenous cartilage transplant with PRP GF (platelet plasma with growth factor) — Arthroscopic reconstruction of cartilage defects in the knee joint using an autogenous PRP GF cartilage transplant.
  Arms: Method of autogenous PRP (Auto Cart-Arthrex) cartilage transplant
Procedure: Arthroscopic reconstruction of the cartilage defects of the knee joint using the microfracture method — Arthroscopic reconstruction of the cartilage defects of the knee joint using the microfracture method.
  Arms: Microfracture method

SUMMARY:
Clinical and comparative evaluation of the treatment results of arthroscopic reconstruction of cartilage defects in the knee joint with the use of autogenous cartilage graft with PRP GF (platelet-rich plasma with growth factors)

DETAILED DESCRIPTION:
The main goal of the research project is to evaluate the results of the treatment of arthroscopic reconstruction of cartilage defects in the knee joint with the use of an autogenous PRP GF cartilage graft. The specific objectives are: to compare the results of treatment of analogous areas of the cartilage defects of the knee joint obtained in the study groups using two methods: microfracture and autogenous PRP GF cartilage graft (Auto Cart-Arthrex method). The results on the operated limb will be compared in both groups both between the groups and with the results of clinical and biomechanical tests on non-operated limbs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years;
* Surgery for ACL damage to the knee joint;
* Arthroscopic surgery;
* No prior knee surgical interventions;
* No additional pathologies in this anatomical area;
* Informed consent of the patient to participate in the study.

Exclusion Criteria:

* Age under 18 or over 65;
* Previous surgical interventions in the examined anatomical area;
* Additional pathologies in this area identified as part of preoperative diagnostics;
* Damage to the second knee joint;
* Failure to comply with the rigor of the same rehabilitation treatment protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-06-22 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | 1 day
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score | 3 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Visual Analogue Score | 6 months after procedure
  Visual Analogue Score - subjective measure for acute and chronic pain. 100-mm VAS ratings of:
  * 0 to 4 mm can be considered no pain;
  * 5 to 44 mm, mild pain;
  * 45 to 74 mm, moderate pain;
  * 75 to 100 mm, severe pain.
Tegner Activity Level Scale (TAS) | 1 day
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS) | 3 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Activity Level Scale (TAS) | 6 months after procedure
  The Tegner Activity Scale (TAS) aims to provide a standardized method in determining the level of activity prior to injury and level of activity post injury that can be documented on a numerical scale.
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.
Tegner Lysholm Knee Scoring Scale | 1 day
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale | 3 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
Tegner Lysholm Knee Scoring Scale | 6 months after procedure
  The Tegner Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
  Grading the Tegner Lysholm Knee Scoring Scale:
  * <65 - poor;
  * 65-83 - fair;
  * 84-90 - good;
  * >90 - excellent.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 1 day
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 3 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
IKDC SUBJECTIVE KNEE EVALUATION FORM | 6 months after procedure
  Interpreted as a measure of function, such that higher scores represent higher levels of function and lower levels of symptoms. A score of 100 is interpreted to mean no limitation with sporting activities or daily living and the complete absence of symptoms.
Body Mass Index (BMI) | 1 day
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 3 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Body Mass Index (BMI) | 6 months after procedure
  BMI is interpreted using standard weight status categories:
  I : below 18.5 kg/m2 - underweight;
  II : 18.5 - 24.9 kg/m2 - healthy weight;
  III : 25.0 - 29.9 kg/m2 - overweight;
  IV : 30.0 kg/m2 and above - obesity.
Magnetic resonance imaging (MRI) | 6 months after procedure
  1,5 Tesli
Ultrasonography (USG) | 6 months after procedure
  Ultrasound examination on the apparatus with the option of elastometry
Biomechanical examination | 3 months after procedure
  On the Biodex 3 System measuring device
Biomechanical examination | 6 months after procedure
  On the Biodex 3 System measuring device

CONTACTS AND LOCATIONS:
Locations (1):
- eMKa MED Medical Center, Wroclaw, Dolnośląsk, Poland

IPD SHARING:
Plan to Share IPD: No